CLINICAL TRIAL: NCT05603741
Title: Local Anesthetic Response in Ehlers-Danlos Syndrome (EDS) and Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB22-1157
Record Dates: First submitted 2022-10-24; First posted 2022-11-03 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Ehlers-Danlos Syndrome; Anesthesia, Local
Keywords: Ehlers-Danlos Syndrome; Local Anesthesia Resistance
MeSH Terms: conditions — Ehlers-Danlos Syndrome | interventions — Sodium Chloride; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Receiving Local Anesthetic Injection (Other): Patients meeting the diagnostic criteria (2017) for Ehlers-Danlos Syndrome
  Healthy control volunteers who do not meet the criteria for Ehlers-Danlos Syndrome
  Interventions: Drug: 0.9% Sodium Chloride Injection; Drug: Lidocaine Injection 2%

INTERVENTIONS:
Drug: 0.9% Sodium Chloride Injection — All participants will be injected subcutaneously with a single 0.5ml dose
  Other Names: Saline
Drug: Lidocaine Injection 2% — All participants will be injected subcutaneously with a single 0.5ml dose
  Other Names: Xylocaine; Lignocaine

SUMMARY:
Local anesthetic resistance is commonly reported by patients with EDS. However, there are no objective data on the occurrence of local anesthetic resistance in EDS patients and in healthy volunteers. The investigators propose to collect such objective data on the frequency of drug resistance and whether any problems with local anesthesia are due to initial ineffectiveness or due to its effects dissipating too soon.

DETAILED DESCRIPTION:
There was a prior large online questionnaire to better understand the issues around local anesthetic resistance. By November 2018, 933 EDS patients (total 1059 respondents) completed the survey, 99.2% of which had previously received local anesthetics. Among these patients, 88% reported that they have "had a problem with local anesthetic injection not working adequately or properly," while only 54% of respondents without EDS reported a similar problem. These data suggests that local anesthetic resistance might be more prevalent in patients with EDS than in the general population. If these findings are true, then this might have significant implications for the appropriate management of these patients during minor surgery and dental procedures.

This study aims to assess the frequency and related issues around local anesthetic resistance in EDS patients, including whether the problem is a lack of analgesia or a timing effect (short duration of action or delayed onset of action), and whether the problem relates only to some local anesthetics or whether there is a problem with the whole class of local anesthetics. This study is completing data originally collected during a 2019 EDS conference.

ELIGIBILITY:
Inclusion Criteria:

* EDS patients, clinically diagnosed hypermobile EDS based on 2017 criteria
* EDS patients with genetically proven non-hypermobile EDS
* Healthy participants, no EDS
* Able and willing to provide informed consent

Exclusion Criteria:

* Known allergy to Lidocaine
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Delta Pain Scores Lidocaine at 5 min [ Time Frame: 5 minutes post-injection ] | 5 minutes post-injection
  Difference between the pain score at the Lidocaine injection locations (compared to a control location) and the saline injection location (compared to a control location). The pain scale is .a 4 level scale from 0 ("absent sensation"), to 1 ("dull pressure"), to 2 ("sharp but less than a control [non-injected] region) to 3 (same or worse than the control region).

SECONDARY OUTCOMES:
Delta Pain Scores Lidocaine at 30 min | 30 minutes post-injection
  Difference between the pain score at the Lidocaine injection locations (compared to a control location) and the saline injection location (compared to a control location). The pain scale is .a 4 level scale from 0 ("absent sensation"), to 1 ("dull pressure"), to 2 ("sharp but less than a control [non-injected] region) to 3 (same or worse than the control region).

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- Cardiovascular Autonomic Research Lab, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No